CLINICAL TRIAL: NCT00755248
Title: Coronary Artery Bypass Grafting: Factors Related to Late Events and Saphenous Graft Patency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Centro Cardiologico Monzino, Centro Cardiologico Monzino
Other Study IDs: BAPPY
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Myocardial Revascularization; Atherosclerosis
Keywords: Coronary Artery Bypass Grafting (CABG); outcome; saphenous graft patency; biochemical factors; genomics
MeSH Terms: conditions — Atherosclerosis | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma,serum, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Pts undergoing CABG or OPCAB
  Interventions: Procedure: Coronary Artery Bypass Grafting

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting — Coronary Artery Bypass Grafting on- or off-pump

SUMMARY:
The purpose of this study is to determine the relations between conventional and unconventional risk factors and adverse clinical events at follow-up (including coronary bypass patency) in patients undergoing surgical myocardial revascularization.

DETAILED DESCRIPTION:
Coronary artery bypass grafting represents one of the most frequent surgical procedure performed in the United States and Europe. The clinical benefit of myocardial revascularization is related to freedom of adverse cardiovascular events and to graft patency, above all of great saphenous vein, which is nowadays the main autologous vessel used for grafting coronaries different from anterior interventricular artery. Unfortunately, phenomena leading to early and, above all, late complications and to graft occlusion are not fully clarified and it so not possible to explain interindividual and temporary variability of progressive stenosis rate only on the basis of classical atherosclerosis risk factors. The aim of our study is to prospectively study the role of conventional risk factors (preoperative risk factors and clinical features) and of unconventional risk factors (genetic polymorphisms, inflammation and coagulation markers) with saphenous late patency and postoperative patients outcome, in particular with regard to adverse clinical events (myocardial infarction, successive stenting procedures, arrhythmias etc.)and to bypass patency.

Plasma venous samples will be collected the day before surgery, at discharge from the hospital, and at follow-up from patients undergoing on-pump and off-pump coronary artery bypass grafting and stored at -80°C; Patients will be followed-up periodically with visits and telephone interviews, and will be also invited to undergo multislice (64 rows) CT scan in order to assess graft patency between 12 and 24 months after surgery.

Finally the relation between conventional and unconventional risk factors with adverse events at follow-up will be assessed with multivariable statistical models.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 to 89
* Elective primary CABG
* Female patients must be non-lactating and not pregnant
* Able and willing to comply with study requirements by signing a consent form

Exclusion criteria

* Concomitant surgery
* Major end organ dysfunction
* Serious intercurrent illness or infection
* Known coagulation disorders
* Emergencies

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-01; Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Parolari, MD, PhD, Principal Investigator — Centro Cardiologico Monzino - Milano
Locations (1):
- Centro Cardiologico Monzino, Milan, Milan, Italy

REFERENCES:
- [Background] 1. American Heart Association. Heart disease and stroke statistics - 2005 update. Dallas, TX: AHA 2004 2. Lytle BW. Prolonging patency - choosing coronary bypass grafts. N Engl J Med 2004; 351: 2262-4 3. Motwani JG et al. Aortocoronary saphenous vein graft disease : pathogenesis, predisposition and prevention. Circulation 1998; 97:916-31 4. Yilmaz M et al. Metabolic syndrome negatively impacts early patency of saphenous vein grafts. Coronary artery disease 2006; 17:41-4 5. Moor E et al. Haemostatic function in patients undergoing coronary artery bypass grafting: perioperative perturbations and relations to saphenous vein graft closure. Thrombosis research 2000; 98:39-49 6. Podgoreanu M et al. New paradigms in cardiovascular medicine. JACC 2005; 46:1965-77 7. Stafford-Smith M et al. Association of genetic polymorphisms with risk of renal injury after coronary bypass graft surgery. Am J Kidney Dusease 2005; 45:519-30 8. Moor E et al. Coagulation factor V (Arg506à Gln) mutation and early saphenous graft occlusion after coronary artery bypass grafting. Thromb Haemost 1998; 80:220-4 9. Yende S et al. Clinical relevance of ACE gene polymorphisms topredict risk of mechanical ventilation after coronary artery bypass surgery. Crit Care Med 2004; 32: 922-27